CLINICAL TRIAL: NCT01609530
Title: Randomized Double Blind Study Comparing Liquid Nitrogen Cryotherapy With Nd:YAG in the Treatment of Verruca Vulgaris
Brief Title: Pulsed 1064nm Nd:YAG in the Treatment of Verruca Vulgaris Versus Conventional Therapy With Liquid Nitrogen Cryotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to accrue the projected number of patients required.
Sponsor: Trinity Health Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSR 11-1215
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Verruca Vulgaris
Keywords: verruca vulgaris; hands; feet; Nd:YAG; laser; cryotherapy
MeSH Terms: conditions — Warts | interventions — Cryotherapy; Heart Rate; Lasers

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trail of standard cryotherapy compared with laser treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: Using sealed envelope assignment, the participant will be placed in study Arm 1 or 2. The investigator will not be masked because the investigator will administer the standard of care cryotherapy or the experimental laser treatment. The outcome assessor will be masked to study group assignment for gathering data from trial participants.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liquid Nitrogen Cryotherapy (Active Comparator): Every two weeks for a total of 5 treatments or until the patient clears, patients in the cryotherapy arm will be treated with 5-7 seconds of freeze time maintaining a 1mm freeze halo around the wart.
  Interventions: Procedure: Liquid Nitrogen Cryotherapy
- Pulsed 1064nm Nd:YAG (Experimental): Every 2 weeks for a total of five treatments or until the wart clears, patients in the laser arm will be treated with the Nd:YAG. The settings will be 180J, 20ms pulse width and 5mm spot size. For warts 3mm or less, a 3mm spot size will be used, 180J and 15ms. If the patient reports no response after treatment, including crusting or blistering, the energy will be increased by 10 J until 200J has been reached.
  Interventions: Procedure: Pulsed 1064nm Nd:YAG

INTERVENTIONS:
Procedure: Liquid Nitrogen Cryotherapy — Every two weeks for a total of 5 treatments or until the patient clears, patients in the cryotherapy arm will be treated with 5-7 seconds of freeze time maintaining a 1mm freeze halo around the wart.
  Other Names: cryotherapy
  Arms: Liquid Nitrogen Cryotherapy
Procedure: Pulsed 1064nm Nd:YAG — Every 2 weeks for a total of five treatments or until the wart clears, patients in the laser arm will be treated with the Nd:YAG. The settings will be 180J, 20ms pulse width and 5mm spot size. For warts 3mm or less, a 3mm spot size will be used, 180J and 15ms. If the patient reports no response after treatment, including crusting or blistering, the energy will be increased by 10 J until 200J has been reached.
  Other Names: laser
  Arms: Pulsed 1064nm Nd:YAG

SUMMARY:
Verruca vulgaris (VV), or the common wart, is a relatively prevalent and often frustrating cutaneous disease to treat. A single, highly effective therapy for the treatment of VV has not been found. Liquid nitrogen is considered the standard of care for VV and studies report a 44% to 47% cure rate. In search of more efficacious and convenient therapeutic options, a variety of lasers have been reported in the treatment of VV including the Nd:YAG laser (1064nm). Lasers offer the potential for decreased treatment associated pain, fewer office visits, higher cure rates and lower recurrence rates. However, many of the available published studies draw conclusions from case reports and small case series without any randomized controlled trials. A randomized, controlled study is needed to evaluate the efficacy of the microsecond Nd:YAG (1064nm) compared to conventional cryotherapy.

This study will use the Cutera CoolGlide Nd:YAG laser that operates in the infrared spectrum at a wavelength of 1064nm. This a single site, double blind, randomized controlled clinical trial to evaluate the efficacy of the Nd:YAG laser (Cutera) in the treatment of verruca vulgaris of the hands and feet versus conventional liquid nitrogen therapy.

The investigators hypothesize that there will be a significantly higher number of warts with complete resolution at 4 months follow-up in the Nd:YAG treated group versus the liquid nitrogen therapy group. The investigators also hypothesize that there will be a faster time to complete resolution of the verruca in the Nd:YAG treated group versus the liquid nitrogen treated group.

DETAILED DESCRIPTION:
Outcome measures: The primary outcome will be complete resolution of the lesion defined as: clinical absence of verruca vulgaris with redevelopment of skin lines on the dorsal surface and dermatoglyphics (ridges of the skin) on the inner surface of the palms and feet, as determined by a blinded clinician investigator blinded to the treatment will evaluate each lesion and determine whether the lesion. A secondary outcome will include: time to complete resolution of the lesion.

2. Objectives and Specific Aims 1.1. Primary objective: To evaluate the efficacy of the Cutera CoolGlide 1064nm Nd:YAG laser in the treatment of verruca vulgaris of the hands and feet versus conventional therapy with liquid nitrogen cryotherapy.

2. Research Design and Methods This a single site double blind (faculty observer and patient blinded; operator/clinician non-blinded), randomized controlled clinical trial to evaluate the efficacy of the Nd:YAG laser (Cutera) in the treatment of verruca vulgaris of the hands and feet versus conventional therapy with liquid nitrogen in 52 patients.

2.2 Study Procedures Informed consent A signed informed consent form will be obtained from each patient prior to entering the study

Physical examination A brief physical examination of the skin including the affected area will be performed. Photographs will be taken of affected areas, prior to and after each treatment from baseline through the fifth treatment follow-up. The investigator will document the number, size and location of each lesion.

Laboratory tests No laboratory testing will be performed for this research project.

Procedure Visit

Initial Visit (DAY 1):

Prior to the clinic visit and treatment:

1. The patient will be screened for inclusion by a study team member using a screening questionnaire (Appendix A).
2. A sub-investigator will review the screening criteria to validate that the patient meets eligibility criteria.
3. Written informed consent will be obtained from the patient before participation in the study (Appendix B).

Treatment 1:

1. The qualifying eligible patient who has consented to participate in the study will be assigned to receive either Nd:YAG laser treatment or liquid nitrogen therapy using a previously established block randomization schema prepared by the research statistician.
2. All lesions will be evaluated and pared with a #15 surgical blade if thickness, a callous, crust or debris is noted, or if hyperkeratosis or other skin thickening is evident which would impede evaluation of the wart.
3. The attending faculty physician will confirm the diagnosis with use a dermatoscope and will be blinded to the treatment assignment.
4. Photos will be taken of the lesions, after paring with a #15 blade to remove any crust or thickened skin above the wart, prior to treatment, and after treatment. A consistent photography procedure (Appendix C) will be used. Each wart will be numbered; size and location will be documented on the Dermatology Study Wart Assessment and Treatment Records (Appendix D). Photographs will be taken before and after treatment.
5. All lesions will be anesthetized with topical lidocaine (LMX 4%) applied under occlusion for 15minutes prior to treatment.
6. All patients will be prepared for treatment in the same manner. They will wear the protective goggles used in laser treatment and will use head phones to muffle the sound of treatment. Both treatment modalities will be turned on prior to the treatment so sounds may not be predictive of the treatment.

8. The patients that have been randomly selected to receive Nd:YAG laser treatment will be fully treated with the following parameters for the laser. If the warts are greater than 3mm the following settings will be used: 20 millisecond pulse width, fluence 180 J/cm2, spot size 5 mm. If warts are 3mm or less in diameter, the laser settings will be: 180 J/cm2, spot size 3mm, pulse width 15 milliseconds. No laser gel will be used during treatment. After each laser pulse, the treated area can be briefly cooled with the tip of the laser. If more than one pulse is needed to cover the entire area of the wart, 10% overlap will be used and area outside of the wart border will not be treated.

9. The patients that have been randomly selected to receive liquid nitrogen treatment will receive liquid nitrogen spray gun for 5-7 seconds creating and maintaining a 1-2 mm freeze halo around lesion for the duration of the application. Use nozzle extender for warts less than 3 mm.

10. Patients will be instructed to avoid treating the warts at home, but they may use vaseline, aquaphor, or plain petrolatum and a band aid as needed for comfort until the next visit .

11. Patients will schedule a return visit in two weeks for assessment of the effects of treatment.

12. Patient treatments will be documented on the appropriate Dermatology Study Wart Treatment Record (Appendix D). Revision of the Dermatology Study Wart Treatment Record is attached with the Request for Revision.

12.1 Document the patient's medications on the Master Medication Record 12.2 Document the patient's warts on the Master Record of Warts

1. Treatments #2, 3, 4, 5 (DAY 14, 28, 42, 56; +/- 7 days) Patient will return at 2week intervals for evaluation and documentation of lesions.
2. An objective faculty observer blinded to treatment, will evaluate wart persistence or clearance at treatments #2, 3, 4, and 5, after the lesion is pared. Faculty will document findings on the Wart Study Attending Faculty Observer Assessment Tool Appendix E).
3. Photos will be taken after paring lesions with a #15 blade; number, size, and location of lesions will be documented, as well as occurrence of any new warts.

   1. If the patient has no clinical lesions present as determined by a blinded faculty clinician, the patient will move on to follow up phase, see below.
   2. If there is still clinical evidence of persisting lesions the patient will be retreated with the same randomized modality as in treatment #1.
   3. If new warts are identified, the investigators will document the number, size, and location of the warts, and photograph the new warts before and after treatment.
   4. Treatment of new warts will be with the same randomized treatment modality to avoid patient un-blinding.
4. All lesions will be anesthetized with topical lidocaine (LMX 4%) applied under occlusion for 15 minutes prior to treatment.
5. All patients will be prepared for treatment in the same manner. They will wear the protective goggles used in laser treatment and will use head phones to muffle the sound of treatment. Both treatment modalities will be turned on prior to the treatment so sounds may not be predictive of the treatment.
6. Proceed with treatment of warts in the same manner as randomization. Complete steps 9- 11 as listed under the initial treatment.

Follow-Up Phase: Clinical Clearance Once a lesion is clinically clear, the patient will move on to the follow up phase. No lesion will be treated more than 5 times. Patients who do not clear after the evaluation of the 5th treatment will be considered treatment failure and will be removed from the study. Patients who fail study treatment will be offered continuing treatment outside of the study through Dermatology Clinic. The patient will be responsible for standard charges for any additional treatment through Dermatology Clinic.

Patients who clear will return to the clinic for evaluation at 1 and 2 months after clinical clearance to determine continued clearance or recurrence. Recurrence will be defined as a new clinical evident lesion that appear in the same location(s) as the previously treated wart(s) up to 2 months post treatment.

1 and 2 Month Follow Up

1. Clinician will perform an examination of the treated areas as in previous visits.
2. Photos will be taken.
3. Size and location of new lesions, if any, will be documented.
4. Recurrence of previously treated lesions will be documented.

4 Month Follow-up

At 4 months following the clearance date, a structured telephone interview will investigate the status of the lesion(s). If the patient is unsure of the status of clearance, the patient will be asked to return for evaluation by the sub-investigator. If the wart recurs or persists, the patient will be offered additional treatment using other options and will be billed for any post-study treatment.

3. Data management and statistical analysis Data Collection and management Data will be collected on paper Case Report forms by the resident physician treating the subject. See data collection tools (Appendix D) and rules in the Procedure Book. Double data entry will be provided by data entry staff into two separate excel spread sheets. Data comparison will be completed by the research statistician. Any discrepancies will be reviewed by the study team. Issues in need of adjudication will be decided by the PI.

Sample size determination: Sample size was calculated based on a formula for effective sample size in a randomized clustered design with binary outcomes. On average, patients will present with approximately three lesions (usually between 1 and 5) requiring treatment. An estimate of a 50% cure rate, using cryotherapy for plantar warts, was drawn from a Cochrane review published in 2006 [10, 11]. We will consider a clinically significant improvement, if at least 80% of the warts treated by Nd:Yag laser are completely resolved at the 6 month visit. We will assume a moderate intra-cluster correlation coefficient of 0.3. Given the cluster design, enrolling 52 patients with, on average, 3 warts each, randomized to one of two treatments, will be needed to provide 84% power to show a statistically significant difference in cure rate. Significance will be set at p<0.05.

Data Management and Analysis All analyses will be done using SAS® 9.2. Demographic and clinical variables will be summarized using means, medians and percentages, as appropriate. To determine whether the primary outcome, complete resolution of each lesion at 2 and 4 months follow-up, is different between treatment groups, we will use a generalized linear mixed model with a binomial distribution, and with initial lesion size and duration, as covariates in the model. The correlation of outcomes within patient will be modeled using a random effect. The secondary outcome, time to complete resolution will be analyzed using a using a multilevel survival model with patient as a random effect and initial lesion size and duration as covariates in the model. To see whether the results are sensitive to missing data, both models will be analyzed with and without the self-reported 4-month outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females, ages 18 - 75
2. Fitzpatrick skin types 1-6
3. Patient is able to read and understand English and will give written informed consent to participate.
4. Patient elects to undergo laser therapy or conventional therapy with liquid nitrogen for the treatment of verruca vulgaris.
5. Clinical evidence of at least one verruca vulgaris, but no more than ten that have not received treatment for at least one month prior to their study start date.
6. Warts to be treated will be located only on the hands or the feet.

Exclusion Criteria:

1. Less than 18 years of age or greater than 75 years of age.
2. Non-English speaking people, who cannot read, understand and sign the consent.
3. Pregnant females.
4. Any form of prior treatment to the area within the last 1 month.
5. Immunosuppressed patients including patients with internal malignancy, on immunosuppressive drugs (including oral steroids), HIV positive or history of connective tissue disease (ie. SLE, DM, Scleroderma).
6. Patients undergoing light therapy including NBUVB, PUVA, high UVB will be excluded from the study until their treatment is complete.
7. Allergy to any components of the topical lidocaine (LMX, 4% lidocaine).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Wart clearance | ~ 6 months
  Patients are treated with either arm of the study every 2 weeks for a total of 10 weeks (5 treatments) or until their warts clear. Patients whose warts clear are then followed up at 1 month and 2 months in person and then at 4 months by phone.

SECONDARY OUTCOMES:
Time to clearance | ~6 months
  Time to clearance will be calculated based on the number of treatments needed to clear the wart.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Auster, MD, Principal Investigator — Saint Joseph Mercy Hospital
Locations (1):
- St. Joseph Mercy Hospital, Ypsilanti, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Tonsy MH, Anbar TE, El-Domyati M, Barakat M. Density of viral particles in pre and post Nd: YAG laser hyperthermia therapy and cryotherapy in plantar warts. Int J Dermatol. 1999 May;38(5):393-8. doi: 10.1046/j.1365-4362.1999.00719.x. PMID 10369554
- [Background] Robson KJ, Cunningham NM, Kruzan KL, Patel DS, Kreiter CD, O'Donnell MJ, Arpey CJ. Pulsed-dye laser versus conventional therapy in the treatment of warts: a prospective randomized trial. J Am Acad Dermatol. 2000 Aug;43(2 Pt 1):275-80. doi: 10.1067/mjd.2000.106365. PMID 10906651
- [Background] Kuykendall-Ivy TD, Johnson SM. Evidence-based review of management of nongenital cutaneous warts. Cutis. 2003 Mar;71(3):213-22. PMID 12661750
- [Background] Park JH, Hwang ES, Kim SN, Kye YC. Er:YAG laser treatment of verrucous epidermal nevi. Dermatol Surg. 2004 Mar;30(3):378-81. doi: 10.1111/j.1524-4725.2004.30104.x. PMID 15008864
- [Background] Tan OT, Hurwitz RM, Stafford TJ. Pulsed dye laser treatment of recalcitrant verrucae: a preliminary report. Lasers Surg Med. 1993;13(1):127-37. doi: 10.1002/lsm.1900130120. PMID 8426521
- [Background] Gooptu C, James MP. Recalcitrant viral warts: results of treatment with the KTP laser. Clin Exp Dermatol. 1999 Mar;24(2):60-3. doi: 10.1046/j.1365-2230.1999.00418.x. PMID 10233653
- [Background] Kopera D. Verrucae vulgares: flashlamp-pumped pulsed dye laser treatment in 134 patients. Int J Dermatol. 2003 Nov;42(11):905-8. doi: 10.1046/j.1365-4362.2003.01994.x. PMID 14636211
- [Background] Han TY, Lee JH, Lee CK, Ahn JY, Seo SJ, Hong CK. Long-pulsed Nd:YAG laser treatment of warts: report on a series of 369 cases. J Korean Med Sci. 2009 Oct;24(5):889-93. doi: 10.3346/jkms.2009.24.5.889. Epub 2009 Sep 23. PMID 19794989
- [Background] Gibbs S, Harvey I. Topical treatments for cutaneous warts. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD001781. doi: 10.1002/14651858.CD001781.pub2. PMID 16855978
- [Background] Killip S, Mahfoud Z, Pearce K. What is an intracluster correlation coefficient? Crucial concepts for primary care researchers. Ann Fam Med. 2004 May-Jun;2(3):204-8. doi: 10.1370/afm.141. PMID 15209195
- [Background] Sterling JC, Handfield-Jones S, Hudson PM; British Association of Dermatologists. Guidelines for the management of cutaneous warts. Br J Dermatol. 2001 Jan;144(1):4-11. doi: 10.1046/j.1365-2133.2001.04066.x. PMID 11167676
- See also: Educational information about warts — http://www.aad.org/skin-conditions/dermatology-a-to-z/warts
- See also: Educational information about warts. — http://emedicine.medscape.com/article/1133317-treatment